CLINICAL TRIAL: NCT06335693
Title: Safety and Efficacy Study of Adjuvant Hypofractionated Radiotherapy Following Radical Prostatectomy for Prostate Cancer
Brief Title: Adjuvant Hypofractionated Radiotherapy for Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhang Huo Jun, Director, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHHHospital
Record Dates: First submitted 2024-03-17; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adjuvant hypofractionated radiotherapy (Experimental): Patients after radical prostatectomy with high-risk pathological factors will receive hypofractionated post-prostatectomy radiotherapy in 15 fractions.
  Interventions: Other: Radiotherapy

INTERVENTIONS:
Other: Radiotherapy — The patients after radical prostatectomy with high-risk pathological factors will receive adjuvant hypofractionated radiation therapy in 15 fractions.

SUMMARY:
Hypofractionated radiation therapy is a new type of radiotherapy which has been shown to play a larger role in the treatment of prostate cancer. The aims of the trial were to evaluate the safety and feasibility of adjuvant hypofractionated radiotherapy following radical prostatectomy for prostate cancer.

DETAILED DESCRIPTION:
The present study will be conducted as a prospective, prospective, single-centre, single-arm clinical trial. Patients after radical prostatectomy with high-risk pathological factors will receive hypofractionated post-prostatectomy radiotherapy in 15 fractions. The primary endpoint of the study is incidence of radiotherapy-related gastrointestinal and genitourinary adverse events,judging by (CTCAE)5.0. The secondary endpoints are progression-free survival (PFS) including biochemical recurrence-free survival (bPFS) and radiological progression-free survival (RPFS), economic evaluations, self-assessment of quality of life including Abbreviated Version of the Expanded Prostate Cancer In-dex Composite Instrument (EPIC-26) and Physical Activity Rank Scale-3 (ARS-3), overall survival (OS) and prostate cancer-specific survival (CSS).

ELIGIBILITY:
Inclusion Criteria:

1. ECOG performance status 0-2.
2. Pathologically confirmed prostate cancer and completion of radical prostatectomy.
3. Postoperative pathological staging pT 3a, pT 3b, pT 4, surgical margins (+) or N1; or serum PSA ≥0.1ng/ml at 6 weeks postoperatively; or serum PSA <0.1ng/ml at 6 weeks postoperatively, with two consecutive persistently elevated PSA (≥0.1ng/ml) without signs of metastasis on clinical imaging (whole-body bone scan (ECT), magnetic resonance imaging (MRI), 68Ga PSMA PET/CT, etc.) .
4. Expected survival time >5 years.
5. Voluntarily accepted this experimental study protocol after being informed of the available treatment options.

Exclusion Criteria:

1. Patients with poor recovery of continence after radical prostatectomy.
2. Patients with a history of pelvic and abdominal radiotherapy.
3. Patients who participated in other clinical trials that were repugnant to the intervention of this trial within 4 weeks prior to the start of this trial.
4. Patients with other malignancies and acute or chronic infections such as human immunodeficiency virus (HIV) (+), hepatitis C virus (HCV) (+) and/or positive syphilis.
5. Patients who are deemed unfit to participate in this clinical trial in the judgement of the investigator, for instance, patients with serious systemic diseases that, in the judgement of the investigator, may interfere with the treatment and evaluation of this trial and its compliance, including serious respiratory, circulatory, neurological, psychiatric, gastrointestinal, endocrine, immunological, urological and other systemic diseases.
6. Patients with radiotherapy-related contraindications.
7. Patients who cannot provide written informed consent and have poor adherence to treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-03-28 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of radiotherapy-related gastrointestinal and genitourinary adverse events | through study completion, an average of 3 years
  Incidence of radiotherapy-related gastrointestinal and genitourinary adverse events

SECONDARY OUTCOMES:
progression-free survival (PFS) | Assessment progression-free survival (PFS) at 3 years
  including biochemical recurrence-free survival (bPFS) and radiological progression-free survival (RPFS)
medical expenses | through study completion, an average of 3 years
  Medical expenses include the cost of examination, hospitalisation, medication, radiation therapy, hospital equipment and any necessary follow-up treatment.
quality of life(QoL) | through study completion, an average of 3 years
  Expanded Prostate Cancer In-dex Composite Instrument 26 (EPIC-26) assesses 26 items in 5 areas, including urinary incontinence, urethral irritation and urethral obstruction symptoms, bowel function, sexual function, sexuality and sex hormone levels. The total score ranges from 0 to 100, with higher scores indicating better quality of life.
overall survival (OS) | Assessment overall survival (OS) at 3 years
  To assess the overall survival (OS)
prostate cancer-specific survival (CSS) | Assessment prostate cancer-specific survival (CSS) at 3 years
  To assess the prostate cancer-specific survival

CONTACTS AND LOCATIONS:
Overall Officials: Huojun Zhang, PhD, Study Director — Changhai Hospital
Locations (1):
- The First Affiliated Hospital of Naval Medical University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data including baseline characteristics,treatment information and follow-up data on toxicity, survival and disease control will be shared.
Supporting Information: Study Protocol
Time Frame: Within 3 years after the publication of the study.
Access Criteria: Data may be shared with radiation oncologists and specialists in surgery who are interested in examining the efficacy and toxicity of hypofractionated radiotherapy following radical prostatectomy. Detailed study protocol should be emailed along with the request of the data. We may carefully review the study protocol, and data will only be shared with well-designed studies.